CLINICAL TRIAL: NCT03685942
Title: Efficacy of Light Therapy Device LUMINETTE® in Major Depressive Disorder(LUMIDEP)
Brief Title: Efficacy of Light Therapy Device LUMINETTE® in Major Depressive Disorder
Acronym: LUMIDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: LUCIMED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIPH 2017-02; IDRCB 2017-A03349-44 (Other: ANSM (French competent authority))
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Unipolar Depression
Keywords: light therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active light therapy (Experimental): Light therapy 1000 lux daily for 30 minutes, as soon as possible after awaking, in preference between 7 and 9 a.m., during 8 weeks in addition to usual treatment
  Interventions: Device: active light therapy (LUMINETTE®)
- placebo light therapy (Placebo Comparator): People receive usual treatment and use a placebo light therapy device (175 lux) daily for 30 minutes, as soon as possible after awaking, in preference between 7 and 9 a.m. during 8 weeks.
  Interventions: Device: placebo light therapy

INTERVENTIONS:
Device: active light therapy (LUMINETTE®) — light therapy on a portable light visor device
  Arms: active light therapy
Device: placebo light therapy — placebo portable light visor device
  Arms: placebo light therapy

SUMMARY:
This study evaluates the addition of light therapy with LUMINETTE device to usual treatment (antidepressant drug and psychotherapy) in the treatment of Major Depressive Disorder (MDD). Half of the participants will receive active light therapy with LUMINETTE device while the other half will receive placebo light therapy with LUMINETTE placebo device.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a world wide spread disorder. According to the World health organization, MDD affects more than 300 million people of all ages in the world. Treatments of MDD include pharmacological treatment and psychotherapy. Pharmacological treatments, mostly serotonin selective reuptake inhibitors, have a delayed onset of action, require long-term treatment and have partial efficacy. In fact, only one third of patients respond to the first antidepressant treatment and two-third after multiple trials. So, there is a need for new treatment strategy.

Light therapy is a well established non pharmacological treatment of seasonal affective disorder, a clinical subtype of affective disorder characterized by recurrent episodes of depression occurring with a seasonal pattern. Patients are exposed to artificial light for a variable duration and intensity. Although the precise mechanism of bright light therapy remains unknown, it is thought to act through the eyes by activating the suprachiasmatic nucleus, the principal circadian pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* MDD diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders I-V (DSM-IV), assessed by means of the Mini Neuropsychiatric International Interview (MINI).
* age between 18 and 60 years.
* affiliation with a welfare scheme.
* complete information on the study received and written informed consent signed

Exclusion Criteria:

* diagnosis of a progressive psychiatric disorder (except MDD and anxiety disorder) according to Axis I of the DSM-IV, assessed by means of the MINI.
* absence of routine care for MDD.
* previous or current LT treatment.
* seasonal affective disorder.
* high suicide risk, assessed by means of the MINI
* ongoing neurological disease.
* retinal pathology.
* participation in another study.
* patient impairment leading to difficulty participating or impossibility or inability to understand the information provided on the study.
* persons cited in Articles L. 1121-5 to L. 1121-8 of the French Public Health Code: pregnant women, parturient or breastfeeding mothers, persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care under duress, persons admitted to a health or social establishment for other goals than research, minors, adults subject to a legal protection, adults who are unable to express their consent and who are not subject to a legal protection measure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg depression rating scale (MADRS) | week 8
  Rating scale measuring depressive symptoms. Each item is scored from 0 to 3, yielding a total between 0 and 27.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | week 8
  Self reported rating scale measuring quality of sleep
Epworth Sleepiness Scale (ESS) | week 8
  Self reported rating scale measuring day time sleepiness
Hamilton Anxiety Rating Scale (HAM-A) | week 8
  Tool measuring the severity of anxiety symptoms.

OTHER OUTCOMES:
electroretinogramm | at inclusion, week 4,8 and 12
  test that measure the functional activity of the retina
Hopkins Verbal Learning Test (HVLT) | week 10
  test of verbal Learning and memory
Montreal Cognitive Assessment (MoCA) | week 10
  screening assessment for detecting cognitive impairment
Stroop test | week 10
  test assessing the ability to inhibit cognitive interference
Trail Making Test (TMT) | week 10
  test evaluating executive functions
Wechsler Adult Intelligence Scale subtest (WAIS) | week 10
  test evaluating memory
optical coherence tomography (OCT) | inclusion and week 12
  evaluation of retinal structure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SCHWITZER, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwitzer T, Le Cam S, Cosker E, Vinsard H, Leguay A, Angioi-Duprez K, Laprevote V, Ranta R, Schwan R, Dorr VL. Retinal electroretinogram features can detect depression state and treatment response in adults: A machine learning approach. J Affect Disord. 2022 Jun 1;306:208-214. doi: 10.1016/j.jad.2022.03.025. Epub 2022 Mar 15. PMID 35301040
- [Derived] Cosker E, Moulard M, Schmitt S, Angioi-Duprez K, Baumann C, Laprevote V, Schwan R, Schwitzer T. Portable light therapy in the treatment of unipolar non-seasonal major depressive disorder: study protocol for the LUMIDEP randomised controlled trial. BMJ Open. 2021 Jul 9;11(7):e049331. doi: 10.1136/bmjopen-2021-049331. PMID 34244279